CLINICAL TRIAL: NCT05505318
Title: Pattern and Outcome of Surgical Treatment of Parotid Gland Neoplasms in Upper Egypt(Retrospective Study)
Brief Title: Pattern and Surgical Treatment of Parotid Gland Neoplasms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Haitham Tharwat Mohamed, Principle investigator, Sohag University
Other Study IDs: soh-med-22-07-17
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Parotid Gland Neoplasm
Keywords: parotid
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- parotid gland neoplasm in upper Egypt

SUMMARY:
in these study we analyze pattern of parotid gland neoplasms according to histopathological types, most common type clinical presentation and type of surgical treatment(superficial parotidectomy or total parotidectomy radical parotidectomy

DETAILED DESCRIPTION:
aim of study is to analyze pattern of parotid glands neoplasms in upper Egypt as regard

1)age 2) sex , 3) clinical presentation :symptom (parotid lump, pain and facial nerve paralysis) and sign (tenderness, fixation of parotid lump and presence of lymph nodes) 4)histopathological types:(benign or malignant 5)surgical options :superficial parotidectomy, total parotidectomy or radical parotidectomy 6)postoperative complications :facial nerve dysfunction, fistula ,recurrence 7) mortality rate all data will be recorded, tabulated , and statistically analyzed .

ELIGIBILITY:
Inclusion Criteria:

* all patient with parotid neoplasm with any age and sex at the period between may2015 to May2021 presented in upper Egypt enrolled in this study all the data will recorded ,tabulated and statistically analyzed emphasizing on:

  1) age. 2)sex. 3)clinical presentation: symptoms (parotid lump ,pain and facial nerve paralysis
  * sign (tenderness ,fixations of parotid lump and presence of lymph nodes) . 4)surgical options : - superficial parotidectomy (partial superficial parotidectomy or formal superficial parotidectomy) .
* total parotidectomy .
* radical parotidectomy. 5)postoperative complications: facial nerve dysfunction, fistula , recurrence) .

  6) mortality rate.

Exclusion criteria:

No exclusion criteria

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: parotid neoplasms patients in upper Egypt
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-05-20 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
pattern of parotid gland neoplasms | after 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Egypt